CLINICAL TRIAL: NCT02052375
Title: A Phase 1, Randomized, Double-Blind, Placebo-Controlled, Multiple-Dose Study To Evaluate the Pharmacokinetics, Pharmacodynamics, Safety and Tolerability of ASP2408 After Subcutaneous Injections in Patients With Rheumatoid Arthritis on Methotrexate
Brief Title: A Study To Evaluate the Pharmacokinetics, Pharmacodynamics, Safety and Tolerability of ASP2408 After Multiple Dose Subcutaneous Injections in Patients With Rheumatoid Arthritis on Methotrexate
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Astellas Pharma Global Development, Inc. (Industry)
Responsible Party: Sponsor
Organization: Astellas Pharma Inc (Industry)
Allocation: Randomized | Model: Parallel | Masking: Quadruple
Other Study IDs: 2408-CL-0201
Record Dates: First submitted 2014-01-30; First posted 2014-02-03 (Estimated); Last update posted 2014-02-06 (Estimated); Status verified 2014-02

CONDITIONS: Rheumatoid Arthritis; Pharmacokinetics of ASP2408
Keywords: Rheumatoid Arthritis; ASP2408; methotrexate
MeSH Terms: conditions — Arthritis, Rheumatoid | interventions — ASP2408

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (4):
- ASP2408 low dosing frequency (Experimental)
  Interventions: Drug: ASP2408
- ASP2408 high dosing frequency (Experimental)
  Interventions: Drug: ASP2408
- Placebo low dosing frequency (Experimental)
  Interventions: Drug: Placebo
- Placebo high dosing frequency (Experimental)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: ASP2408 — subcutaneous injection
  Arms: ASP2408 high dosing frequency; ASP2408 low dosing frequency
Drug: Placebo — subcutaneous injection
  Arms: Placebo high dosing frequency; Placebo low dosing frequency

SUMMARY:
The purpose of this study is to assess the safety, tolerability and pharmacokinetics (PK) of two dosing regimens of multiple, subcutaneous (sc) injections of ASP2408 in patients with Rheumatoid Arthritis (RA) on Methotrexate (MTX) and to evaluate the pharmacodynamics (PD) of ASP2408.

DETAILED DESCRIPTION:
This is an ascending dose frequency study. There are two cohorts of active and placebo patients. The first cohort is dosed every 4 weeks for a total of 3 doses. The second cohort is dosed every two weeks for a total of 3 doses.

ELIGIBILITY:
Inclusion Criteria:

* Subject weighs at least 50 kg.
* Subject has a body mass index (BMI) of ≤ 35 kg/m2.
* Subject's 12-lead electrocardiogram (ECG) results are normal at Screening and Day 1 prior to study drug dosing or, if abnormal, the abnormality is not clinically significant as determined by the Investigator.
* Subject has Rheumatoid Arthritis (RA) that was diagnosed according to the 1987 revised criteria of the American College of Rheumatology (ACR) ≥ 6 months prior to Screening.
* Subject meets the ACR 1991 revised criteria for Global Functional Status in RA, Class I, II or III at Screening.
* Subject MUST be on concomitant methotrexate (MTX):

  * for ≥ 3 months prior to Day 1, AND
  * at a stable dose (10 - 25 mg/week) for ≥ 28 days prior to Day 1 and throughout the study.
* Subject's other related medications taken for the treatment of RA at the time of Screening must meet the noted stability requirements and remain on a stable regimen, as follows:

  * Non-steroidal anti-inflammatory drugs (NSAIDs), selective cyclooxy-genase-2 (COX-2) inhibitors, oral corticosteroids (≤ 10 mg of prednisone, or equivalent, daily) or low dose opioids (≤ 30 mg of oral morphine, or equivalent, daily) must be stable for ≥ 28 days prior to Screening and remain so throughout the Treatment and Observation Period.
* Hydroxychloroquine (Plaquenil®) and sulfasalazine must have started ≥ 2 months, and be stable for ≥ 28 days, prior to Day 1.

Exclusion Criteria:

* Subject has an ongoing infection or has had an infection requiring intravenous antibiotics within 1 month prior to Day 1.
* Subject has a past history of serious opportunistic infection.
* Subject has a positive Mantoux tuberculin skin or QuantiFERON-TB Gold test within 90 days of, or at Screening, and has not completed an adequate course of antimicrobial therapy per CDC guidelines.
* Subject received any live or live-attenuated vaccine within 30 days prior to Day 1.
* Subject received any of the following:

  * Anakinra (Kineret®), etanercept (Enbrel®), or adalimumab (Humira®) within 60 days prior to Day 1.
  * Rituximab (Rituxan®) or any other anti-CD20 antibody within 180 days prior to Day 1.
  * Leflunomide (Arava®) within 60 days prior to drug dosing on Day 1, unless the subject has undergone cholestyramine washout at least 30 days prior to Day 1.
  * Oral or injectable gold, azathioprine, penicillamine, cyclosporine, or tacrolimus within 30 days prior to Day 1.
  * Cyclophosphamide within 180 days prior to Day 1.
* Subject has received any CTLA4-Ig molecule (including, but not limited to abatacept [Orencia®] and belatacept [Nulojix]).
* Subject has participated in a previous clinical study with treatment with ASP2408 or ASP2409 or has participated in another dose cohort of the current trial.
* Subject has previously participated in any interventional clinical study, or has received an experimental agent within 56 days or 5 half-lives, whichever is longer, prior to Day 1.
* Subject has a history of prolonged QT syndrome.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2012-06; Primary Completion 2013-12 (Actual); Study Completion 2013-12 (Actual)

PRIMARY OUTCOMES:
Pharmacokinetic parameter of ASP2408: AUCtau | Days 1, 2, 3, 4, 5, 6, 8, 10, 15, 22, 36, 38, 43, 50, 57, 66, 71, 78, 85, 113, 141
  Area Under the Concentration-Time curve for a dosing interval (AUCtau)
Pharmacokinetic parameter of ASP2408: Cmax | Days 1, 2, 3, 4, 5, 6, 8, 10, 15, 22, 36, 38, 43, 50, 57, 66, 71, 78, 85, 113, 141
  Maximum Concentration (Cmax)
Pharmacokinetic parameter of ASP2408: Tmax | Days 1, 2 ,3, 4, 5, 6, 8, 10, 15, 22, 36, 38, 43, 50, 57, 66, 71, 78, 85, 113, 141
  Time to Attain Cmax (Tmax)
Pharmacokinetic parameter of ASP2408: Ctrough | Days 1, 2, 3, 4, 5, 6, 8, 10, 15, 22, 36, 38, 43, 50, 57, 66, 71, 78, 85, 113, 141
  Trough Concentration (Ctrough)
Safety assessed by adverse events (AEs), laboratory tests, electrocardiograms (ECGs), physical examinations, pulse oximetry, vital signs and Anti-ASP2408 antibody (ADA) formulation | Up to 1 year

SECONDARY OUTCOMES:
Composite of pharmacokinetics of ASP2408: t1/2, Vz/F, CL/F, | Days 1, 2, 3, 4, 5, 6, 8, 10, 15, 22, 36, 38, 43, 50, 57, 66, 71, 78, 85, 113, 141
  Apparent Terminal Elimination Half-life (t1/2), Volume of distribution (Vz/F), Apparent Body Clearance (CL/F)
Pharmacodynamic parameter of ASP2408: CD86 receptor occupancy | Days 1, 2, 3, 4, 5, 6, 8, 10, 15, 22,36, 38, 43, 50, 57, 66, 71, 72, 78, 85,113, 141
  Cluster of Differentiation 86, a co-stimulatory ligand on antigen-presenting cells; alternate notation for B7.2 (CD86)

CONTACTS AND LOCATIONS:
Overall Officials: Senior Medical Director, Study Director — Astellas Pharma Global Development, Inc.
Locations (3):
- United States (3):
  - Pinnacle Research Group, LLC, Anniston, Alabama
  - Altoona Center for Clinical Research, Duncansville, Pennsylvania
  - Metroplex Clinical Research Center, LLC, Dallas, Texas